CLINICAL TRIAL: NCT01371864
Title: Families and Pediatric Cardiac Surgery Multidisciplinary Teams: How Well Do We Communicate?
Brief Title: Families and Pediatric Cardiac Surgery Multidisciplinary Teams: How Well Do We Communicate
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1772; UNCDRE (Other Grant/Funding Number: University of North Carolina Department of Anesthesiology)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2013-03

CONDITIONS: Communication
Keywords: Congenital cardiac disease; Teamwork; Communication; Peri-operative
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pediatric Cardiothoracic Team: This group consists of members of the cardiothoracic surgery team: The attending physician, the fellow physician, the nurses, and the physician assistants.
- Critical Care Team: This group consists of the nurses and physicians who work in the pediatric intensive care unit and the neonatal intensive care unit caring for patients who require cardiothoracic surgery.
- Subspecialty Team: This group consists of physicians and nurses from pediatric cardiology and pediatric anesthesiology who care for children who require cardiothoracic surgery.
- Parent: This group consists of the parent or legal guardian of the pediatric patient who requires cardiothoracic surgery.

SUMMARY:
Purpose:

-To evaluate the peri-operative communication between families and the pediatric cardiac surgery team.

Method:

-In this study the investigators plan to utilize structured interview and survey of parents/legal guardians and health care providers of children undergoing cardiac surgery in the United States of America.

DETAILED DESCRIPTION:
Every day clinicians face challenges when attempting to negotiate their way through dialogues with families whose children require surgical intervention in the near future. The area of clinician-patient communication with pediatric families is under-researched and highlights a pressing clinical problem. There are several adult studies that describe the content and nature of patient-physician communications at the time of cardiac surgery. However, there are no studies that evaluate the communications between nursing, physicians, and pediatric patient's families at the time of cardiac surgery. Further knowledge in this area is valuable in that a disparity between the these groups can lead to medical error, damage the clinician-patient relationship and provide grounds for dissatisfaction, complaints, or claim. This research will provide insight into what patient's families value in their communications with the medical team and assist the medical community in better meeting our children's families needs.

ELIGIBILITY:
Inclusion Criteria:

* Primary language is English
* > 18 years age
* Nurse, physician, physician assistant, or parent / legal guardian of a pediatric patient who requires cardiothoracic surgery at the North Carolina Children's Hospital.

Exclusion Criteria:

* Primary language is not English. The interviewers all speak English as their primary language. People whose primary language is other than English will only be excluded if they do not have the ability to converse in English with the interviewers.
* <18 years of age. The parent / legal guardian must be of age to be the primary caregiver able to make decisions for their child.
* People with an intellectual or mental impairment that prohibits their capacity to make medical decisions for their child. Our research aims to investigate the relationship between the parent / legal guardians of pediatric cardiac surgery patients who interact with the pediatric cardiac surgery multidisciplinary team. These individuals must have sufficient mental capacity to be able to provide consent for their child to undergo surgery. Individuals with intellectual or mental impairment that prohibits their ability to give consent are therefore excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from a tertiary care academic children's hospital including:
  * Inpatient population within the pediatric critical care unit, neonatal critical care unit, and the cardiac intermediate care unit.
  * Outpatient population including the pediatric cardiothoracic surgery clinic patients.
  * Hospital personnel
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Peri-operative risk information | 1 week
  Parental and provider assessment of the content and nature of communications in the peri-operative time period. Specifically, the quantity and type of risk information required before consenting for surgery.

SECONDARY OUTCOMES:
Informed decisions | 1 week
  Parental and provider assessment of the content and nature of communications in the peri-operative time period. Specifically, the family's ability to make informed decisions.
Trust in the medical team | 1 week
  Parental and provider assessment of the content and nature of communications in the peri-operative time period. Specifically, the families trust in the medical team.
Desire for disclosure of peri-operative complications | 1 week
  Parental and provider assessment of the content and nature of communications in the peri-operative time period. Specifically, families desire for disclosure of peri-operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Cherissa C Hanson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States